CLINICAL TRIAL: NCT02424877
Title: Cell Phone Based Automated Monitoring of Patients With Early Rheumatoid Arthritis
Acronym: SandRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medcare Oy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SandRA-WI177026
Record Dates: First submitted 2015-04-20; First posted 2015-04-23 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; drug treatment; compliance; outcome
MeSH Terms: conditions — Arthritis, Rheumatoid; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SandRA (Experimental): cell phone monitoring
  Interventions: Procedure: SandRA
- Control (No Intervention): conventional monitoring

INTERVENTIONS:
Procedure: SandRA — SandRA software sends SMS messages to a patient asking questions about the usage and adverse effects of prescribed drugs and about the severity of rheumatoid arthritis. The answer messages are interpreted automatically.
  Arms: SandRA

SUMMARY:
The purpose of this study is to determine whether automated remote monitoring of patients with early rheumatoid arthritis by the SandRA software and short message service of cell phones increases patient compliance and helps to identify patients needing re-assessment of medication before scheduled visits. This might result in better clinical outcome and cost-effectiveness.

DETAILED DESCRIPTION:
To improve monitoring of patients with early RA the investigators have developed an automated remote monitoring system SandRA (Showing-any-need-for-Re-Assessment) based on short message service (SMS) of cell phones and patients' global assessment of the severity of RA (PtGA) on a numeric scale of 0 to 10.

SandRA software sends every 2 to 6 weeks automatically an SMS to a patient's cell phone, and the patient answers by one push on keyboard. The patients' answers are recorded in SandRA and automatically analysed. If answers indicate non-adherence, adverse events, or missed target, the system automatically sends SMS: "Your nurse will call you within 2 work days", and the nurse gets an alarm by e-mail. If needed, an extra visit is arranged for treatment adjustment.

Preliminary studies show that PtGA given by cell phone has sufficient convergent validity. Structured feedback from patients has been favourable and most professionals assess the system as feasible.

The objective of this study is to investigate the impact of SandRA monitoring on clinical outcomes of RA, on patients' quality of life and drug adherence, as well as consumed resources. Cost-effectiveness of SandRa is estimated.

Methods Consecutive incident patients (200) with RA are enrolled. Those, who can use SMS messages of cell phone, who understand the SandRA system, and are willing, are included. After informed consent the patients are randomized into two groups: 1) SandRA group and 2) control group.

The patients randomized into SandRA group are instructed as usual. Regular doctor visits are scheduled at 3 months and at 6 months, when the SandRa monitoring ends. The following clinical data will be gathered. 1) ACR core data set at baseline, at 3 and 6 months, and at possible extra visits; 2) radiographs of the hands and the feet at baseline (if not taken within 6 months); 3) antirheumatic medication and the possible causes of switches and changes over the 6 months 4) patient confidence (VAS) at each doctor visit; 5) quality of life (SF-36) at baseline and at 6 months. Patient feedback of the system by a structured questionnaire is gathered at 6 months.

The patients in the control group are treated as usual. Follow-up visits are scheduled as needed. The same clinical data as in SandRA group are collected at baseline and at 6 months.

In the both groups concomitant diseases and medications as well as age, sex, and education level are recorded at baseline. The consumption of resources is assessed as the number of contacts (doctor visits, nurse visits, as well as phone calls scheduled and non-scheduled) with the outpatient clinic over the 6-month follow-up.

In addition, the patients are assessed at 12 months, when the ACR Core Data Set is gathered.

The radiographs at baseline and ACR Core Data Set at doctor visits, safety laboratory tests, and assessment visits at 3, 6, and 12 months are included in the normal clinical care. No extra visits are required because of the study.

ELIGIBILITY:
Inclusion Criteria:

* Fulfillment of the EULAR 2010 classification criteria for rheumatoid arthritis
* Commencement of the first anti rheumatic medication
* Ability to use short message service of cell phones,
* Comprehension of the function of the SandRA monitoring system
* Willingness to participate.

Exclusion Criteria:

- Failure to fulfill the inclusion criteria.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2016-01-30 (Actual); Study Completion 2017-01-02 (Actual)

PRIMARY OUTCOMES:
remission | at 6 months (co-primary 12 months)
  number of remissions at each arm, defined by no tender or swollen joints (44 joints) and normal CRP

SECONDARY OUTCOMES:
patient confidence | at 0, 3, and 6 months
  visual analogue scale
quality of life | at 0, 3, and 6 months
  SF-36
drug adherence | during 6 months
  stoppage of drugs, adverse events
consumption of resources | during 6 months
  extra phone calls, extra visits

CONTACTS AND LOCATIONS:
Overall Officials: Kari Puolakka, MD, PhD, Principal Investigator — South Carelia Central Hospital
Locations (2):
- Finland (2):
  - Central Finland Central Hospital, Jyväskylä
  - South Karelia Central Hospital, Lappeenranta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mottonen T, Hannonen P, Leirisalo-Repo M, Nissila M, Kautiainen H, Korpela M, Laasonen L, Julkunen H, Luukkainen R, Vuori K, Paimela L, Blafield H, Hakala M, Ilva K, Yli-Kerttula U, Puolakka K, Jarvinen P, Hakola M, Piirainen H, Ahonen J, Palvimaki I, Forsberg S, Koota K, Friman C. Comparison of combination therapy with single-drug therapy in early rheumatoid arthritis: a randomised trial. FIN-RACo trial group. Lancet. 1999 May 8;353(9164):1568-73. doi: 10.1016/s0140-6736(98)08513-4. PMID 10334255
- [Background] Grigor C, Capell H, Stirling A, McMahon AD, Lock P, Vallance R, Kincaid W, Porter D. Effect of a treatment strategy of tight control for rheumatoid arthritis (the TICORA study): a single-blind randomised controlled trial. Lancet. 2004 Jul 17-23;364(9430):263-9. doi: 10.1016/S0140-6736(04)16676-2. PMID 15262104
- [Background] Brus H, van de Laar M, Taal E, Rasker J, Wiegman O. Determinants of compliance with medication in patients with rheumatoid arthritis: the importance of self-efficacy expectations. Patient Educ Couns. 1999 Jan;36(1):57-64. doi: 10.1016/s0738-3991(98)00087-1. PMID 10036560
- [Background] Schoels M, Kapral T, Stamm T, Smolen JS, Aletaha D. Step-up combination versus switching of non-biological disease-modifying antirheumatic drugs in rheumatoid arthritis: results from a retrospective observational study. Ann Rheum Dis. 2007 Aug;66(8):1059-65. doi: 10.1136/ard.2006.061820. Epub 2007 Feb 16. PMID 17307765
- [Background] Rohekar G, Pope J. Test-retest reliability of patient global assessment and physician global assessment in rheumatoid arthritis. J Rheumatol. 2009 Oct;36(10):2178-82. doi: 10.3899/jrheum.090084. Epub 2009 Sep 15. PMID 19755617
- [Background] Pincus T, Bergman M, Sokka T, Roth J, Swearingen C, Yazici Y. Visual analog scales in formats other than a 10 centimeter horizontal line to assess pain and other clinical data. J Rheumatol. 2008 Aug;35(8):1550-8. Epub 2008 Jun 15. PMID 18597409
- [Derived] Kuusalo L, Sokka-Isler T, Kautiainen H, Ekman P, Kauppi MJ, Pirila L, Rannio T, Uutela T, Yli-Kerttula T, Puolakka K; SandRA Study Group. Automated Text Message-Enhanced Monitoring Versus Routine Monitoring in Early Rheumatoid Arthritis: A Randomized Trial. Arthritis Care Res (Hoboken). 2020 Mar;72(3):319-325. doi: 10.1002/acr.23846. PMID 30740935